CLINICAL TRIAL: NCT04087317
Title: Comparison Between 2 Pain Analgesic Protocols Following Vaginal Delivery
Brief Title: Vaginal Postpartum Pain Management Protocol Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Gal Bachar MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rambam Health Care Center.
Record Dates: First submitted 2019-08-07; First posted 2019-09-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pain; Post Partum Depression; Opioid Use; Breast Feeding
MeSH Terms: conditions — Pain; Depression, Postpartum; Breast Feeding | interventions — Acetaminophen; Tablets; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Women following a vaginal delivery, with no exclusion criteria to participate in the study, will be addressed. After receiving all the information about the study, women who choose to participate will be consented.
  All participants will be randomized to either scheduled analgesic administration (study group) or analgesic administration per women's request (control group) as accustomed at the investigator's unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed time interval group. (Experimental): Patients received oral 1-gram paracetamol and 400 milligram ibuprofen every 6 hours, in the first 24 hours postpartum. After 24 hours postpartum and until discharge, they will receive analgesics at maternal request. At any time, if a woman experienced pain despite the prescribed treatment, the next line of treatment was MIR (morphine immediate release, 10 mg tablet).
  Interventions: Drug: Paracetamol 1000 Mg Oral Tablet; Drug: Ibuprofen 400Mg Tab; Drug: MIR
- 'On-demand' group. (Experimental): Patients received oral 1-gram paracetamol and 400 milligram ibuprofen at maternal request. At any time, if a woman experienced pain despite the prescribed treatment, the next line of treatment was MIR (morphine immediate release, 10 mg tablet).
  Interventions: Drug: Paracetamol 1000 Mg Oral Tablet; Drug: Ibuprofen 400 mg; Drug: MIR

INTERVENTIONS:
Drug: Paracetamol 1000 Mg Oral Tablet — The drug will be administrated when the woman arrive to the maternity unit, and every 6 hours thereafter, for first 24 hours following delivery.
  Other Names: Acetaminophen
  Arms: Fixed time interval group.
Drug: Ibuprofen 400Mg Tab — The drug will be administrated when the woman arrive to the maternity unit, and every 6 hours thereafter, for first 24 hours following delivery.
  Arms: Fixed time interval group.
Drug: Paracetamol 1000 Mg Oral Tablet — The drug will be administrated after a maternal request, by at least 6 hours apart between dosages.
  Other Names: Acetaminophen
  Arms: 'On-demand' group.
Drug: Ibuprofen 400 mg — The drug will be administrated after a maternal request, by at least 6 hours apart between dosages.
  Arms: 'On-demand' group.
Drug: MIR — At any time, if a woman experienced pain despite the prescribed treatment, the next line of treatment was MIR (morphine immediate release, 10 mg tablet).

SUMMARY:
Untreated postpartum pain has been associated with increased risk of opioid use, postpartum depression and development of persistent pain. In this study the investigators will investigate whether a scheduled administration of analgesics is superior to administration of analgesics based on patient request following a vaginal delivery.

DETAILED DESCRIPTION:
More than two million women deliver vaginally every year in the United States (US). Along with the joy and happiness of having a new member in the family, women may suffer from cramping pain and lower abdomen discomfort following uterine involution; perineal pain due to perineal trauma or episiotomy; and nipple pain from breastfeeding or breast engorgement.

A stepwise approach using multimodal combination of medications can effectively provide an individualized pain management for women in their postpartum period. The first step includes non-opioid analgesics (as paracetamol and NSAIDs), step two adds milder opioids (as codeine, tramadol and oral morphine), and step three incorporates stronger opioids (as parenteral morphine).

In this study the investigators will investigate whether a scheduled administration of analgesics is superior to administration of analgesics based on patient request following a vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Women following term vaginal delivery.

Exclusion Criteria:

1. Under Age 18 years or older than 45 years.
2. Women with chronic pain syndrome.
3. Women with relative or absolute contraindications for paracetamol or NSAIDs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) score difference in the 24 first hours. | In the first 24 hours postpartum.
  Pain control using visual analog scale (VAS) score of 0 (no pain/ least satisfaction) to 10 (worst pain/ highest satisfaction).

SECONDARY OUTCOMES:
Amount of additional analgesia requirements. | Up to maternal discharge (5 days)
  Total amount of additional analgesia up to maternal discharge.
Total analgesia requirements. | Up to 48 hours postpartum.
  Total amount of analgesics use during 48 hours following a vaginal delivery.
Breastfeeding rate. | Up to 48 hours postpartum.
  The rate of women who breastfeed their newborns and breastfeeding frequency.
Treatments side effects. | Up to 48 hours postpartum.
  Side effects reported by the medical staff (clinically or laboratory) or women receiving analgesia.
Visual analog scale (VAS) score difference up to maternal discharge. | At any time, if a woman experienced pain despite the prescribed treatment, the next line of treatment was MIR (morphine immediate release, 10 mg tablet). up to 5 days.
  Pain control using visual analog scale (VAS) score of 0 (no pain/ least satisfaction) to 10 (worst pain/ highest satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Gal Bachar, MD, Principal Investigator — Rambam Medical Health Center
Locations (1):
- Rambam, Ramat Yishai, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bachar G, Alter A, Justman N, Buchnik Fater G, Farago N, Ben-David C, Abu-Rass H, Siegler Y, Hajaj A, Landau-Levin M, Zipori Y, Khatib N, Weiner Z, Vitner D. Fixed-time interval vs on-demand oral analgesia after vaginal delivery: a randomized controlled trial. Am J Obstet Gynecol MFM. 2024 May;6(5):101372. doi: 10.1016/j.ajogmf.2024.101372. Epub 2024 Apr 5. PMID 38583715
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388